CLINICAL TRIAL: NCT02380326
Title: Innovation in Endobronchial Sampling : Integration of Virtual Bronchoscopic Navigation in the Current Diagnostic Algorithm and the Use of Micro-CT for Tissue Analysis
Brief Title: Innovation in Endobronchial Sampling
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Yserbyt Jonas, MD, KU Leuven
Other Study IDs: 150302V02
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Diffuse Interstitial Lung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — transbronchial biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung transplant recipients: Lung transplant recipients with diffuse parenchymal abnormalities subjected to advanced endoscopic imaging modalities
  Interventions: Procedure: Advanced endoscopic imaging modalities
- Diffuse intersitial lung disease: Patients suffering from diffuse intersitial lung disease without a certain diagnosis subjected to advanced endoscopic imaging modalities
  Interventions: Procedure: Advanced endoscopic imaging modalities

INTERVENTIONS:
Procedure: Advanced endoscopic imaging modalities — Virtual bronchoscopic navigation, confocal laser endomicroscopy, micro CT

SUMMARY:
Evaluating an integrated diagnostic work-up of virtual navigation bronchoscopy (VNB), confocal laser endomicroscopy and micro computerized tomography (micro-CT) in the diagnostic path of pulmonary lesions in the non-oncological patient.

DETAILED DESCRIPTION:
The region(s) of interest that has/have to be sampled, will be selected upfront. Guided by the endobronchial pathway that is created by virtual bronchoscopy, the flexible bronchoscope will be navigated to the regions of interest and an optical biopsy of the region will be obtained using pCLE. One biopsy sample will be processed in the endoscopy suite to be able to prepare it for micro-CT analysis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of diffuse pulmonary disease necessitating bronchoscopic evaluation.
* Informed consent available
* Age > 18
* FVC > 50%pred
* DLCO > 35%pred
* PaO2 > 55 mmHg, pCO2 < 45 mmHg (ambient air)
* No exclusion criteria

Exclusion Criteria:

* Age > 75
* Systolic arterial pressure in the pulmonary artery : PAPS >40mmHg
* Platelet count <100000/µl
* INR > 1.4
* BMI >30
* Diffuse bullous lung disease
* Active anti-platelet or anticoagulant treatment
* Active heart failure or unstable coronary heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients and diffuse interstitial lung disease without certain diagnosis
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | postprocedural

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Yserbyt, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium